CLINICAL TRIAL: NCT05951582
Title: The Effect of Plyometric Exercises on Physical Fitness and Technical Skills of Football Players
Brief Title: The Effects of Plyometric on Physical Fitness and Technical Skills of Football Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/01413 Asim Abdul Rehman
Record Dates: First submitted 2023-07-07; First posted 2023-07-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Physical Fitness and Technical Skills
Keywords: Plyometrics, physical fitness, technical skill and football.
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Plyometrics) (Experimental): This group will receive 8 weeks of upper and lower body plyometric exercises protocol. The session will last for 60 minutes and 3 time per week. 1-minute rest period is there between each exercise and each repetition and 3-5 minute for each set.
  Interventions: Other: Plyometric Exercises
- Group B (Conventional) (Experimental): This group will receive 8 weeks of upper and lower body strength exercises protocol. The session will last for 60 minutes and 3 times per week.
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Plyometric Exercises — The group will receive plyometric exercises in a controlled environment. Following Plyometrics were performed.
  1. Horizontal jumps over hurdle.
  2. Standing long jump
  3. Front cone hops
  4. Forward-backward run
  5. Double leg horizontal jump
  6. Lateral jump over hurdle
  7. Side to side sprint
  8. Jumps over low hurdles
  9. Split squat jump
  10. Cone hops with change of sprint direction
  11. Lateral jump over hurdle
  12. Side to side slide and hops.
  13. Lateral and horizontal jump
  14. Cone hops with 180o turn
  15. Vertical, Lateral, and horizontal jump
  16. Lateral cone jump
  17. Single leg lateral jump
  18. Diagonal Jumps.
  19. Standing long jump with diagonal sprint.
  20. Single leg vertical jump
  21. Cone hop with 1800 turn
  22. Skipping over cone
  Arms: Group A (Plyometrics)
Other: Conventional Exercises — The group will receive conventional exercises in a controlled environment. Following conventional exercises were performed.
  1. Single Leg Squat/ Lunges
  2. Modified Box Step Ups
  3. Press Ups
  4. Box Jumps
  5. Shoulder Press
  6. Standing Band Row
  7. Band Butterfly Pills
  Arms: Group B (Conventional)

SUMMARY:
This study aimed to assess the effectiveness of plyometric exercises on the physical fitness and technical skills of football players in Quetta, Baluchistan

DETAILED DESCRIPTION:
Football (soccer) is a popular sport that is played both competitively and recreationally. It is acknowledged as a repeated exercise involving both aerobic and anaerobic metabolic systems (Beato et al., 2018). Youth are especially passionate about the sport (Di Salvo et al., 2006), being the fourth most popular sport for females in high schools and the fifth most popular sport for men (Brown, 2014). Football players spend the most of their time on the pitch, where there is a high risk of injury because it is a contact sport. Football players need to be both physically and mentally fit to manage the tremendous demands of the game, which call for exceptional levels of memory, planning, focus, and other mental abilities. On the other hand, having good balance is necessary for both a successful sporting career and the prevention of musculoskeletal injuries. (Sheppard & Young, 2006) Plyometric, also known as jump training, has gained significant recognition as a valuable training method for enhancing physical fitness and technical skills in football players. This specialized form of exercise involves explosive movements that activate fast-twitch muscle fibers, which are essential for producing the quick bursts of power required for running, jumping, and changing directions during game-play (Slimani, Chamari, Miarka, Del Vecchio, & Chéour, 2016). Plyometric workouts promote muscular growth and boost the ability to maintain high-intensity activities throughout a match because they put the muscles through repeated, powerful contractions. Football players can sustain their optimum performance level. Plyometric workouts require precise body control and coordination, which directly translate to improved balance and agility on the pitch. These abilities are necessary for football players to move through crowded spaces, evade opponents, and perform challenging maneuvers with grace (Markovic & Mikulic, 2010).

Athletes can use plyometric workouts to develop their lower-body strength, power, coordination, and agility. Examples include horizontal jumps over hurdles, standing long jumps, split squat jumps, diagonal jumps, 180-degree cone hops, and sprints while skipping. Athletes can thrive in sports that involve quick changes in direction by using these workouts, which are created to stress particular muscle groups and movement patterns. (Behm & Chaouachi, 2011)Plyometric exercise promotes agility which is crucial skill, allowing them to change direction rapidly while maintaining control and balance, by improving neuromuscular coordination and muscular power, leading to quicker and more precise movement execution. (Miller et al., 2006)Exercises such as lateral bounds, cone drills, and ladder drills are commonly used in plyometric training to enhance agility (Markovic & Mikulic, 2010).

Football players are more formidable in both offensive and defensive situations because to plyometric activities that boost the legs' explosive power and vertical leap. Football players who have improved their agility, balance, and jumping skills have a competitive advantage that allows them to excel in key situations and dramatically advance their team's chances of winning. (Faude, Koch, & Meyer, 2012) Plyometric training simulates these demands by promoting the development of fast-twitch muscle fibers, increasing reactive strength, and improving the ability to produce force quickly (Slimani et al., 2016). Additionally, plyometric exercises deliver an SSTS (sport-specific training stimulus) that closely mimics the motions made on a football pitch. Rather than taking a broad view of physical fitness and technical football skills, most previous study has focused on individual physical fitness components such as power or speed(Little, Williams, & Research, 2005). More research is needed to fully comprehend the impact of plyometric training on various aspects of physical fitness and technical football ability. Previous studies did not fully comprehend the potential benefits of plyometric training on football players' overall performance. That 'why this study is conducted to evaluate the effects of plyometric on physical as well technical skill among football players.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  1. Male football player
  2. Age between 18-32 years

Exclusion Criteria:

Participant failing to fall in this category would be excluded of the study.

1. History of metabolic diseases.
2. History of recent fractures.
3. History of trauma / injury in last month

Ages: 18 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Anaerobic Endurance | 8 weeks
  The 300 Yard Shuttle Test is used to test of anaerobic endurance, in which the participants run 25 yards and back, repeating this for 12 runs of 25 yards (300 yard total), changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Lower Extrmity Strength | 8 weeks
  The vertical jump test is to check the strength of the lower extremity, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
3-hop test (Lower Extrimity Power) | 8 weeks
  To test the explosive leg power, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Aerobic Fitness | 8 weeks
  The Yo-Yo Intermittent Tests the participants have a short active break (5 and 10 seconds for the intermittent endurance and intermittent recovery test, respectively), changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Speed and Agility | 8 weeks
  For speed, acceleration and agility training of the athlete The Run-a-Three Test is fitness test that assesses both speed and agility. The run-a-three involves sprinting over the actual pitch distance three times, incorporating two 180 degree turns. This test not only assesses speed, but also technique on the turn and running the bat in at the end, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Agility | 8 weeks
  The 505 Agility test is a test of 180 degree turning ability. The test may also be adapted for specific testing by having the subject dribble a soccer ball, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Ability to control and manipulate the ball using their head | 8 weeks
  Head ball juggling tests in soccer players are commonly used to assess and develop specific skills related to heading the ball. The number of consecutive headers or the time a player can keep the ball in the air using only their head can provide insights into their heading proficiency and coordination, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Instep Juglling the Football Skill | 8 weeks
  To check the instep skill of football players, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Footbal Driblling Skills | 8 weeks
  To check dribble in tight space, control, speed and agility. The figure 8 dribbling test in soccer is a drill designed to assess a player's dribbling skills, agility, and control of the ball while maneuvering through a set course, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
ability to maintain control of the ball while dribbling | 8 weeks
  The controlled speed dribbling test in soccer is a drill designed to assess a player's ability to maintain control of the ball while dribbling at a controlled and consistent speed. It evaluates their ball control, touch, coordination, and decision-making skills, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Passing and receiving accuracy | 8 weeks
  The passing and receiving test in soccer is a drill designed to assess a player's passing accuracy, technique, communication, and ability to receive a pass effectively. It focuses on the fundamental skills required for successful passing and receiving in a game scenario, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Ability to Generate Power and Accuracy | 8 weeks
  The power shooting test in soccer is a drill designed to assess a player's ability to generate power and accuracy in their shooting technique. It focuses on evaluating a player's shooting strength, technique, and ability to strike the ball with power and precision, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.
Ability to Execute Accurate and Powerful Long-Distance Passes | 8 weeks
  The driven long ball test in soccer is a drill used to evaluate a player's ability to execute accurate and powerful long-distance passes with speed and precision. It focuses on assessing their technique, decision-making, and execution of driven passes over extended distances, changes from the Baseline, 2nd week, 4th week, 6th week and 8th week will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar A Awan, PhD, Principal Investigator — Faculty of Rehabilitation & Allied Health Sciences, Riphah International University; Asim A Rehman, DPT, Principal Investigator — Rehabilitation Department, Shaikh Muhammad Bin Zayyed Al-Nahyan Institute of Cardiology, Quetta, Balochistan, Pakistan
Locations (1):
- Rehabilitation Department, Sheikh Muhammad bin Zayyed Al-Nahyan Institute of Cardiology, Quetta, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beato M, Bianchi M, Coratella G, Merlini M, Drust B. Effects of Plyometric and Directional Training on Speed and Jump Performance in Elite Youth Soccer Players. J Strength Cond Res. 2018 Feb;32(2):289-296. doi: 10.1519/JSC.0000000000002371. PMID 29176387
- [Background] Di Salvo V, Baron R, Tschan H, Calderon Montero FJ, Bachl N, Pigozzi F. Performance characteristics according to playing position in elite soccer. Int J Sports Med. 2007 Mar;28(3):222-7. doi: 10.1055/s-2006-924294. Epub 2006 Oct 6. PMID 17024626
- [Background] Sheppard JM, Young WB. Agility literature review: classifications, training and testing. J Sports Sci. 2006 Sep;24(9):919-32. doi: 10.1080/02640410500457109. PMID 16882626
- [Background] Spurrs RW, Murphy AJ, Watsford ML. The effect of plyometric training on distance running performance. Eur J Appl Physiol. 2003 Mar;89(1):1-7. doi: 10.1007/s00421-002-0741-y. Epub 2002 Dec 24. PMID 12627298
- [Background] Markovic G, Jukic I, Milanovic D, Metikos D. Effects of sprint and plyometric training on muscle function and athletic performance. J Strength Cond Res. 2007 May;21(2):543-9. doi: 10.1519/R-19535.1. PMID 17530960
- [Background] Ramirez-Campillo R, Meylan C, Alvarez C, Henriquez-Olguin C, Martinez C, Canas-Jamett R, Andrade DC, Izquierdo M. Effects of in-season low-volume high-intensity plyometric training on explosive actions and endurance of young soccer players. J Strength Cond Res. 2014 May;28(5):1335-42. doi: 10.1519/JSC.0000000000000284. PMID 24751658
- [Background] Behm DG, Chaouachi A. A review of the acute effects of static and dynamic stretching on performance. Eur J Appl Physiol. 2011 Nov;111(11):2633-51. doi: 10.1007/s00421-011-1879-2. Epub 2011 Mar 4. PMID 21373870
- [Background] Miller MG, Herniman JJ, Ricard MD, Cheatham CC, Michael TJ. The effects of a 6-week plyometric training program on agility. J Sports Sci Med. 2006 Sep 1;5(3):459-65. eCollection 2006. PMID 24353464
- [Background] Markovic G, Mikulic P. Neuro-musculoskeletal and performance adaptations to lower-extremity plyometric training. Sports Med. 2010 Oct 1;40(10):859-95. doi: 10.2165/11318370-000000000-00000. PMID 20836583
- [Background] Ramirez-Campillo R, Gallardo F, Henriquez-Olguin C, Meylan CM, Martinez C, Alvarez C, Caniuqueo A, Cadore EL, Izquierdo M. Effect of Vertical, Horizontal, and Combined Plyometric Training on Explosive, Balance, and Endurance Performance of Young Soccer Players. J Strength Cond Res. 2015 Jul;29(7):1784-95. doi: 10.1519/JSC.0000000000000827. PMID 25559903
- [Background] Faude O, Koch T, Meyer T. Straight sprinting is the most frequent action in goal situations in professional football. J Sports Sci. 2012;30(7):625-31. doi: 10.1080/02640414.2012.665940. Epub 2012 Mar 6. PMID 22394328
- [Background] Slimani M, Chamari K, Miarka B, Del Vecchio FB, Cheour F. Effects of Plyometric Training on Physical Fitness in Team Sport Athletes: A Systematic Review. J Hum Kinet. 2016 Oct 14;53:231-247. doi: 10.1515/hukin-2016-0026. eCollection 2016 Dec 1. PMID 28149427
- [Background] Sheppard JM, Young WB, Doyle TL, Sheppard TA, Newton RU. An evaluation of a new test of reactive agility and its relationship to sprint speed and change of direction speed. J Sci Med Sport. 2006 Aug;9(4):342-9. doi: 10.1016/j.jsams.2006.05.019. Epub 2006 Jul 17. PMID 16844413
- [Background] Faude O, Roth R, Di Giovine D, Zahner L, Donath L. Combined strength and power training in high-level amateur football during the competitive season: a randomised-controlled trial. J Sports Sci. 2013;31(13):1460-7. doi: 10.1080/02640414.2013.796065. Epub 2013 Jun 17. PMID 23768214
- [Background] Little T, Williams AG. Specificity of acceleration, maximum speed, and agility in professional soccer players. J Strength Cond Res. 2005 Feb;19(1):76-8. doi: 10.1519/14253.1. PMID 15705049
- [Background] Ometto L, Vasconcellos FV, Cunha FA, Teoldo I, Souza CRB, Dutra MB, et al. How manipulating task constraints in small-sided and conditioned games shapes emergence of individual and collective tactical behaviours in football: A systematic review. 2018;13(6):1200-14.
- [Background] Bin Shamshuddin MH, Hasan H, Azli MS, Mohamed MN, Razak FAAJIJoHM, Sciences S. Effects of plyometric training on speed and agility among recreational football players. 2020;8(5).
- [Background] Spiteri T, Nimphius S, Hart NH, Specos C, Sheppard JM, Newton RU. Contribution of strength characteristics to change of direction and agility performance in female basketball athletes. J Strength Cond Res. 2014 Sep;28(9):2415-23. doi: 10.1519/JSC.0000000000000547. PMID 24875426
- [Background] Thomas K, French D, Hayes PR. The effect of two plyometric training techniques on muscular power and agility in youth soccer players. J Strength Cond Res. 2009 Jan;23(1):332-5. doi: 10.1519/JSC.0b013e318183a01a. PMID 19002073
- [Background] Saez-Saez de Villarreal E, Requena B, Newton RU. Does plyometric training improve strength performance? A meta-analysis. J Sci Med Sport. 2010 Sep;13(5):513-22. doi: 10.1016/j.jsams.2009.08.005. Epub 2009 Nov 7. PMID 19897415
- [Background] Gharah, B. E. (2017). The effect of plyometric training on agility and balance. Journal of Physical Education and Sport, 17(3), 1086-1090.
- [Background] Gabbett TJ, Kelly JN, Sheppard JM. Speed, change of direction speed, and reactive agility of rugby league players. J Strength Cond Res. 2008 Jan;22(1):174-81. doi: 10.1519/JSC.0b013e31815ef700. PMID 18296972
- [Background] Kean CO, Behm DG, Young WB. Fixed foot balance training increases rectus femoris activation during landing and jump height in recreationally active women. J Sports Sci Med. 2006 Mar 1;5(1):138-48. eCollection 2006. PMID 24198691
- [Background] Ramirez-Campillo R, Alvarez C, Henriquez-Olguin C, Baez EB, Martinez C, Andrade DC, Izquierdo M. Effects of plyometric training on endurance and explosive strength performance in competitive middle- and long-distance runners. J Strength Cond Res. 2014 Jan;28(1):97-104. doi: 10.1519/JSC.0b013e3182a1f44c. PMID 23838975
- [Background] Thomas C, Jones PA, Rothwell J, Chiang CY, Comfort P. An Investigation Into the Relationship Between Maximum Isometric Strength and Vertical Jump Performance. J Strength Cond Res. 2015 Aug;29(8):2176-85. doi: 10.1519/JSC.0000000000000866. PMID 25647649
- [Background] Brown FF. The Influence of Sex, Training Status, and Fatty Acid Supplementation on T-lymphocyte Populations at Rest and in Response to Acute Exercise. 2014.